CLINICAL TRIAL: NCT00014534
Title: Phase III Study Comparing Sequential Chemotherapy (AG-ITP) To Cisplatin And Gemcitabine As Adjuvant Treatment After Cystectomy For Transitional Cell Carcinoma Of The Bladder
Brief Title: Combination Chemotherapy in Treating Patients With Bladder Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-90104; P30CA008748 (NIH); CALGB-90104; MSKCC-00138; NCI-G01-1935; CDR0000068554 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2001-04-10; First posted 2003-06-10 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-07

CONDITIONS: Bladder Cancer
Keywords: stage III bladder cancer; stage IV bladder cancer; transitional cell carcinoma of the bladder
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Filgrastim; Cisplatin; Doxorubicin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gemcitabine + cisplatin (Active Comparator)
  Interventions: Drug: cisplatin; Drug: gemcitabine hydrochloride
- Gemcitabine + Doxorubicin + Pegfilgrastim (Active Comparator)
  Interventions: Biological: filgrastim; Drug: doxorubicin hydrochloride; Drug: gemcitabine hydrochloride

INTERVENTIONS:
Biological: filgrastim — 6 mg sub Q
  Arms: Gemcitabine + Doxorubicin + Pegfilgrastim
Drug: cisplatin — 60 mg/sq m IV
  Arms: Gemcitabine + cisplatin
Drug: doxorubicin hydrochloride — 50 mg/ sq m IV
  Arms: Gemcitabine + Doxorubicin + Pegfilgrastim
Drug: gemcitabine hydrochloride — 1000 mg/ sq m IV for Gem + cis arm and 2000 mg/sq m IV for gem + dox + peg arm

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Randomized phase III trial to compare different combination chemotherapy regimens in treating patients who have advanced bladder cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the survival of patients with completely resected locally advanced transitional cell carcinoma of the bladder treated with adjuvant doxorubicin and gemcitabine followed by paclitaxel and cisplatin vs adjuvant cisplatin and gemcitabine.

Secondary

* Compare the toxicity profiles of these regimens in these patients.

OUTLINE: This is a randomized study. Patients are stratified according to primary tumor status (<T4 vs T4), number of positive lymph nodes (0 or unknown vs 1-5 vs >5), and number of dissected nodes (0-10 or unknown vs > 10). Patients are randomized to one of two treatment arms.

* Arm I: Patients receive adjuvant gemcitabine IV over 30 minutes on days 1, 8, and 15 and cisplatin IV over 30-60 minutes on day 1. Treatment repeats every 4 weeks for up to 4 courses in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive adjuvant doxorubicin IV over 45 minutes followed by gemcitabine IV over 2 hours on day 1. Patients also receive filgrastim (G-CSF) subcutaneously (SC) daily on days 3-10. Treatment repeats every 14 days for up to 4 courses in the absence of disease progression or unacceptable toxicity. Beginning 14 days after the completion of doxorubicin and gemcitabine, patients receive paclitaxel IV over 3 hours and cisplatin IV over 20-30 minutes on day 1. Patients also receive G-CSF SC daily on days 3-10 or 4-11. Treatment repeats every 14 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 18 months, every 6 months for 18 months, and then annually thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed transitional cell carcinoma of the bladder

  * Any T, N+, M0 OR
  * T3a-4a, N0, M0
* At least 6 weeks but no more than 3 months since prior complete resection of bladder

  * Cystoprostatectomy plus pelvic lymph node dissection in males
  * Cystectomy/total abdominal hysterectomy/bilateral salpingo-oophorectomy plus pelvic lymph node dissection in females
  * Negative surgical margins
* Carcinoma in situ allowed
* No partial cystectomy or transurethral bladder tumor resection as definitive loco-regional therapy
* Prostate cancer detected in resected specimen allowed if post-operative PSA is no more than 0.05 mg/dL
* No metastatic or recurrent disease by post-operative chest x-ray and CT scan of abdomen and pelvis

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-1

Hematopoietic:

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 150,000/mm^3

Hepatic:

* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 2 times ULN
* AST ≤ 2 times ULN

Renal:

* Creatinine ≤ 1.5 mg/dL OR
* Creatinine clearance ≥ 60 mL/min

Cardiovascular:

* Normal cardiac function by history, physical exam, or chest radiograph
* Left ventricular ejection fraction at least 50% by radionuclide ventriculogram or echocardiogram, for prior cardiac disease
* No New York Heart Association class III or IV heart disease
* No serious cardiac arrhythmias including first-, second-, and third-degree heart block

Other:

* Negative pregnancy test
* No uncontrolled infection
* No other active cancer within the past 5 years except non-melanoma skin cancer or curatively treated carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior systemic chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior radiotherapy to bladder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2004-03; Primary Completion 2005-07 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Overall survival | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Dean Bajorin, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (285):
- United States (285):
  - CCOP - Mayo Clinic Scottsdale Oncology Program, Scottsdale, Arizona
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Arroyo Grande Community Hospital, Arroyo Grande, California
  - Rebecca and John Moores UCSD Cancer Center, San Diego, California
  - Kaiser Permanente Medical Office -Vandever Medical Office, San Diego, California
  - Veterans Affairs Medical Center - San Diego, San Diego, California
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - Veterans Affairs Medical Center - San Francisco, San Francisco, California
  - Aurora Presbyterian Hospital, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose Cancer Center at Penrose Hospital, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Presbyterian - St. Luke's Medical Center, Denver, Colorado
  - St. Joseph Hospital, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - CCOP - Colorado Cancer Research Program, Incorporated, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Front Range Cancer Specialists, Fort Collins, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Hope Cancer Care Center at Longmont United Hospital, Longmont, Colorado
  - St. Mary-Corwin Regional Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thorton, Colorado
  - Beebe Medical Center, Lewes, Delaware
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - St. Francis Hospital, Wilmington, Delaware
  - Lombardi Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Lynn Regional Cancer Center of Boca Raton Community Hospital, Boca Raton, Florida
  - Michael & Dianne Bienes Comprehensive Cancer Center at Holy Cross Hospital, Fort Lauderdale, Florida
  - Memorial Cancer Institute at Memorial Regional Hospital, Hollywood, Florida
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Ella Milbank Foshay Cancer Center at Jupiter Medical Center, Jupiter, Florida
  - Watson Clinic, Lakeland, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Phoebe Cancer Center at Phoebe Putney Memorial Hospital, Albany, Georgia
  - Emory University Hospital - Atlanta, Altanta, Georgia
  - Hematology and Oncology of Northeast Georgia, Athens, Georgia
  - MBCCOP-Medical College of Georgia Cancer Center, Augusta, Georgia
  - John B. Amos Community Cancer Center, Columbus, Georgia
  - Curtis & Elizabeth Anderson Cancer Institute at Memorial Health University Medical Center, Savannah, Georgia
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Louis A. Weiss Memorial Hospital, Chicago, Illinois
  - Eureka Hospital, Eureka, Illinois
  - Galesburg Clinic, Galesburg, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - InterCommunity Cancer Center of Western Illinois, Galesburg, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hopedale Medical Complex, Hopedale, Illinois
  - Joliet Oncology Hematology Associates, Limited - West, Joliet, Illinois
  - Provena St. Mary's Wasser Regional Cancer Center - Kankakee, Kankakee, Illinois
  - Kewanee Hospital, Kewanee, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology/Hematology Associates of Central Illinois, P.C., Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - St. Margaret's Hospital, Spring Valley, Illinois
  - Valley Cancer Center, Spring Valley, Illinois
  - Regional Cancer Center at Memorial Medical Center, Springfield, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - St. Francis Hospital and Health Centers, Beech Grove, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Indiana University Cancer Center, Indianapolis, Indiana
  - William N. Wishard Memorial Hospital, Indianapolis, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - Saint Joseph Regional Medical Center - Plymouth Campus, Plymouth, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - McFarland Clinic, P.C., Ames, Iowa
  - St. Luke's Hospital, Cedar Rapids, Iowa
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Mercy Cancer Center at Mercy Medical Center, Cedar Rapids, Iowa
  - Genesis Regional Cancer Center at Genesis Medical Center, Davenport, Iowa
  - Genesis Medical Center - West Campus, Davenport, Iowa
  - Mercy Capitol Hospital, Des Moines, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Wendt Regional Cancer Center at Finley Hospital, Dubuque, Iowa
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Siouxland Hematology-Oncology Associates, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Medical Oncology and Hematology Associates - West Des Moines, West Des Moines, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, P.A. - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Kingman, Kingman, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Cancer Center of Kansas, P.A. - Parsons, Parsons, Kansas
  - Pratt Cancer Center of Kansas, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates in Womens Health, Wichita, Kansas
  - Cancer Center of Kansas, P.A., Wichita, Kansas
  - Cancer Center of Kansas, P.A. - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Central Maine Medical Center, Lewiston, Maine
  - Maine Center for Cancer Medicine and Blood Disorders - Scarborough, Scarborough, Maine
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Union Hospital Cancer Center at Union Hospital, Elkton MD, Maryland
  - Lawrence Memorial Hospital of Medford, Medford, Massachusetts
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Borgess Medical Center, Kalamazooaa, Michigan
  - William Beaumont Hospital - Royal Oak Campus, Royal Oak, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Mercy and Unity Hospitals, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Meeker County Memorial Hospital, Litchfield, Minnesota
  - St. John's Hospital, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - Veterans Affairs Medical Center - Minneapolis, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Medical Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Clinic, Saint Louis Park, Minnesota
  - Cancer Care Center at Regions Hospital, Saint Paul, Minnesota
  - St. Joseph's Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Cancer Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Woodwinds Hospital, Woodbury, Minnesota
  - Missouri Cancer Associates, Columbia, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - St. Anthony's Cancer Center, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Deaconess Billings Clinic - Downtown, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare, Billings, Montana
  - Deaconess Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - St. James Community Hospital, Butte, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Sletten Regional Cancer Institute, Great Falls, Montana
  - St. Peter's Hospital, Helena, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Eastern Montana Cancer Center, Miles City, Montana
  - Community Medical Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Cancer Institute of New Jersey at the Cooper University Hospital, Camden, New Jersey
  - Veterans Affairs Medical Center - East Orange, East Orange, New Jersey
  - CCOP - Northern New Jersey, Hackensack, New Jersey
  - Cancer Institute of New Jersey at Hamilton, Hamilton, New Jersey
  - Fox Chase Virtua Health Cancer Program - Marlton, Marlton, New Jersey
  - Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Fox Chase Virtua Health Cancer Program at Virtua West Jersey, Voorhees Township, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Charles R. Wood Cancer Center at Glens Falls Hospital, Glens Falls, New York
  - Lipson Cancer and Blood Center at Rochester General Hospital, Rochester, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Long Island Cancer Center at Stony Brook University Hospital, Stony Brook, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., Syracuse, New York
  - Veterans Affairs Medical Center - Syracuse, Syracuse, New York
  - Community General Hospital of Greater Syracuse, Syracuse, New York
  - Randolph Hospital, Asheboro, North Carolina
  - Batte Cancer Center at Northeast Medical Center, Concord, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - John Smith, Jr./Dalton McMichael Cancer Center at Morehead Memorial Hospital, Eden, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Moses Cone Regional Cancer Center at Wesley Long Community Hospital, Greensboro, North Carolina
  - Lenoir Memorial Cancer Center, Kinston, North Carolina
  - Annie Penn Cancer Center, Reidsville, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Wilson Medical Center, Wilson, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Medcenter One Health System, Bismarck, North Dakota
  - Mid Dakota Clinic, P.C., Bismarck, North Dakota
  - St. Alexius Medical Center, Bismarck, North Dakota
  - Akron City Hospital at Summa Health System, Akron, Ohio
  - St. Elizabeth Boardman Cancer Center, Boardman, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Ireland Cancer Center at University Hospitals of Cleveland and Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University, Columbus, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Riverside Cancer Services, Columbus, Ohio
  - Mount Carmel West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Community Oncology Group - Independence, Independence, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Middletown Regional Hospital, Middletown, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - Mercy Medical Center Oncology Unit, Springfield, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - St. Joseph Health Care Center, Warren, Ohio
  - Mount Carmel Cancer Services at Mount Carmel St. Ann's Hospital, Westerville, Ohio
  - Cleveland Clinic - Wooster, Wooster, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - St. Elizabeth Cancer Center at St. Elizabeth Health Center - Youngstown, Youngstown, Ohio
  - Genesis - Good Samaritan Hospital, Zanesville, Ohio
  - Oklahoma University Medical Center, Oklahoma City, Oklahoma
  - Legacy Mount Hood Medical Center, Glesham, Oregon
  - Cancer Treatment Center at Merle West Medical Center, Klamath Falls, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Comprehensive Cancer Center at Legacy Good Samaritan Hospital & Medical Center, Portland, Oregon
  - Providence Cancer Center at Providence Portland Medical Center, Portland, Oregon
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Institute of Oncology at Vilnius University, Portland, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Central Pennsylvania Hematology and Medical Oncology Associates, PC, Lemoyne, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Riddle Memorial Hospital, Media, Pennsylvania
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Joan Karnell Cancer Center at Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Hillman Cancer Center at University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Pottstown Memorial Regional Cancer Center, Pottstown, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Miriam Hospital at Lifespan, Providence, Rhode Island
  - Rose Ramer Cancer Clinic at Anderson Area Medical Center, Anderson, South Carolina
  - Roper St. Francis Healthcare - Roper Hospital, Charleston, South Carolina
  - Bon Secours St. Francis Health System, Greenville, South Carolina
  - Greenville Hospital System Cancer Center, Greenville, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Sioux Valley Hospital and University of South Dakota Medical Center, Sioux Falls, South Dakota
  - Avera McKennan Hospital and University Health Center, Sioux Falls, South Dakota
  - Medical X-Ray Center, Sioux Falls, South Dakota
  - Vanderbilt-Ingram Cancer Center at Vanderbilt Medical Center, Nashville, Tennessee
  - Danville Regional Medical Center, Danville, Virginia
  - Providence Cancer Center at Sacred Heart Medical Center, Spokane, Washington
  - Providence Cancer Center at Holy Family Hospital, Spokane, Washington
  - Cancer Center at Southwest Washington Medical Center, Vancouver, Washington
  - West Virginia University - Robert C. Byrd Health Sciences Center - Charleston Division, Charleston, West Virginia
  - St. Mary's Medical Center, Huntington, West Virginia
  - Mary Babb Randolph Cancer Center at West Virginia University Hospitals, Morgantown, West Virginia
  - Fox Valley Hematology and Oncology, Appleton, Wisconsin
  - Gundersen Lutheran Cancer Center at Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - UW Health Oncology, Madison, Wisconsin
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin
  - University of Wisconsin Cancer Center at Aspirus Wausau Hospital, Wausau, Wisconsin
  - Welch Cancer Center, Sheridan, Wyoming